CLINICAL TRIAL: NCT07157007
Title: A Multicenter, Open-Label, Randomized Phase 2a Study to Evaluate Safety and Efficacy of Ratutrelvir and Standard of Care in Non-hospitalized Symptomatic Adult Participants With Mild to Moderate COVID-19
Brief Title: Early-stage Trial to Determine a Safe and Effective Dose for Ratutrelvir in Patients With Mild to Moderate COVID-19
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Traws Pharma, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 83-0060-0002
Record Dates: First submitted 2025-09-03; First posted 2025-09-05 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2026-01

CONDITIONS: COVID - 19
MeSH Terms: conditions — COVID-19 | interventions — nirmatrelvir and ritonavir drug combination

STUDY DESIGN:
Intervention Model Description: Participants will be randomized into 3 study arms (30 participant per arm) to receive study drug and standard of care therapy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Ratutrelvir (83-0060) non-randomised (Experimental)
  Interventions: Drug: Ratutrelvir (83-0060) non-randomised
- Paxlovid (Active Comparator): Standard of care
  Interventions: Drug: Paxlovid
- Ratutrelvir (83-0060) (Experimental)
  Interventions: Drug: Ratutrelvir (83-0060)

INTERVENTIONS:
Drug: Ratutrelvir (83-0060) non-randomised — 83-0060, a covalent inhibitor of the SARS-CoV-2 main protease (Mpro; 3CL)
  Arms: Ratutrelvir (83-0060) non-randomised
Drug: Paxlovid — Paxlovid (Nirmatrelvir+ Ritonavir , boosted 3CL-protease inhibitor)
  Arms: Paxlovid
Drug: Ratutrelvir (83-0060) — 83-0060, a covalent inhibitor of the SARS-CoV-2 main protease (Mpro; 3CL)
  Arms: Ratutrelvir (83-0060)

SUMMARY:
This is an Early-stage Clinical Trial to Determine a Safe and Effective Dose for Ratutrelvir in Patients With Mild to Moderate COVID-19. It will also learn about the safety of drug Ratutrelvir. Participants will take a study drug as well as a standard therapy. A descriptive statistics will be used to present the study results.

DETAILED DESCRIPTION:
This is a multicenter, open-label, randomized Phase 2a study to evaluate the safety and efficacy of 83-0060 (Ratutrelvir) and Nirmatrelvir-Ritonavir (Paxlovid) in non-hospitalized symptomatic adult participants with mild to moderate COVID-19.

ELIGIBILITY:
Inclusion Criteria:

1. Confirmed SARS-CoV-2 infection for 120 h prior to randomization.
2. Initial onset of signs/symptoms attributable to COVID-19 within 5 days prior to randomization.
3. At least one of the symptoms attributable to COVID-19 present within 24 hours prior to the Day 1 with the severity score of 1 or higher according to the following scoring system for the assessment of severity of:

Exclusion Criteria:

Medical Conditions:

1. History, current need for hospitalization or anticipated need for hospitalization for the medical treatment of COVID-19.
2. Urgent or expected need for nasal high-flow oxygen therapy or positive pressure ventilation, invasive mechanical ventilation or ECMO.
3. Known medical history of active liver disease .
4. Receiving dialysis or history of moderate to severe renal impairment.
5. Compromised immune system.
6. Acute episode of chronic respiratory diseases, including bronchial asthma, chronic obstructive pulmonary disease within 30 days before screening.
7. Suspected or confirmed concurrent active systemic infection..

   Prior/Concomitant Therapy:
8. Has received or is expected to receive any dose of a SARS-CoV-2 vaccine within 4 months of screening and during the participation in the study.
9. Concomitant use of any medications or substances that are strong inducers of CYP3A4

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-09-16 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Safety based on adverse events incidence | 28 days
  Adverse events incidence will be described using descriptive statistics methods
Safety based on adverse events severity | 28 days
  Adverse events severity will be assessed by current version of CTCAE

SECONDARY OUTCOMES:
Efficacy based on Time (days) to sustained recovery of all targeted COVID-19 signs/symptoms through Day 28 | 28 days
Efficacy based on Time to sustained recovery of each targeted COVID-19 symptom through Day 28. | 28 days
PK characteristics of 83-0060 based on Maximum Plasma Concentration (Cmax) | 11 days
PK characteristics of 83-0060 based on Area under the concentration time curve from 0 to time of last quantifiable concentration (AUClast) | 11 days
PK characteristics of 83-0060 based on Time to Cmax ( Tmax) | 11 days

CONTACTS AND LOCATIONS:
Locations (15):
- Australia (4):
  - Novatrial, Charlestown, New South Wales
  - Key Health, Sydney, New South Wales
  - Momentum Clinical Research Taringa, Brisbane, Queensland
  - Paratus Clinical(Clinical Trials Institute, Torquay), Torquay, Victoria
- South Korea (5):
  - Chonnam National University Hospital, Gwangju, Donggu
  - The Catholic University of Korea, Eunpyeong St. Mary's Hospital, Seoul, Eunpyeong-gu
  - Wonju Severance Christian Hospital, Wŏnju, Gangwon-do
  - Inha University Hospital, Incheon, Jung-gu
  - Hallym University Sacred Heart Hospital Gangnam, Seoul, Seoul
- Taiwan (5):
  - Kaohsiung Medical University Hospital, Kaohsiung City, Kaohsiung
  - Taichung Veterans General Hospital, Taichung, Taichung
  - Taipei Medical University Hospital, Taipei, Taipei
  - Taoyuan General Hospital, Taoyuan District, Taoyuan
  - Chang Gung Memorial Hospital, Linkou Branch, Taoyuan District, Taoyuan
- Research Institute of Virology, Tashkent, Tashkent, Uzbekistan

IPD SHARING:
Plan to Share IPD: No